CLINICAL TRIAL: NCT03553875
Title: Memantine for the Treatment of Social Deficits in Youth With Disorders of Impaired Social Interactions: A Randomized-controlled Trial
Brief Title: Memantine for the Treatment of Social Deficits in Youth With Disorders of Impaired Social Interactions
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: put on hold by the IRB
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gagan Joshi, Director, Autism Spectrum Disorder Program in Pediatric Psychopharmacology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018P001082
Record Dates: First submitted 2018-06-01; First posted 2018-06-12 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Autism; Autism Spectrum Disorder; Nonverbal Learning Disability
Keywords: Autism; Massachusetts General Hospital
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; non-verbal learning disabilities | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Memantine (Active Comparator): Memantine administered in tablet form twice daily titrated to a maximum dose of 20 mg for 12 weeks.
  Interventions: Drug: Memantine Hydrochloride
- Placebo (Placebo Comparator): Subjects in the placebo control group will receive a matched placebo pill with no active ingredients. This will be administered twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine Hydrochloride — Participating children and adolescents with Non-Verbal Learning Disorder and related conditions (NVLD-RC) who meet the eligibility criteria will be randomly assigned to memantine for the course of the 12-week randomized controlled trial (RCT).
  Arms: Memantine
Drug: Placebo — Participating children and adolescents with Non-Verbal Learning Disorder and related conditions (NVLD-RC) who meet the eligibility criteria will be randomly assigned to placebo for the course of the 12-week randomized controlled trial (RCT).
  Arms: Placebo

SUMMARY:
This study is a 12-week randomized-controlled trial of memantine hydrochloride (Namenda) for the treatment of social impairment in youth with Non-Verbal Learning Disorder, High-Functioning Autism Spectrum Disorder, and related conditions. Eligible participants will be males and females ages 8-18.

This study consists of up to 6 visits to Massachusetts General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Male & female subjects ages 8-18 years (inclusive).
* Diagnostic Statistical Manual (DSM)-5 Autism Spectrum Disorder (ASD) diagnostic criteria as established by clinical diagnostic interview
* At least moderate severity of social impairment as measured by a total raw score of ≥85 on the parent/guardian-completed Social Responsiveness Scale-Second Edition (SRS-2)14 and a score of ≥4 on the clinician-administered Clinical Global Impression-Severity scale (CGI-S)17.

Exclusion Criteria:

* IQ ≤70 based on the Wechsler Abbreviated Scale of Intelligence-II (WASI-II) Vocabulary and Matrix Reasoning subtests
* Impaired communicative speech
* Subjects currently treated with the following medications (known to impact glutamate levels): Lamotrigine, Amantadine, N-acetylcysteine, D-cycloserine
* Subjects treated with a psychotropic medication not listed above on a dose that has not been stable for at least 4 weeks prior to study baseline.
* Co-administration of drugs that compete with memantine for renal elimination using the same renal cationic system, including hydrochlorothiazide, triamterene, metformin, cimetidine, ranitidine, quinidine, and nicotine
* Initiation of a new psychosocial intervention within 30 days prior to randomization.
* Subjects who are pregnant and/or nursing.
* Subjects with a history of non-febrile seizures without a clear and resolved etiology.
* Subjects with a history of or a current liver or kidney disease.
* Clinically unstable psychiatric conditions or judged to be at serious suicidal risk.
* Subjects who meet on the Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS-E) for alcohol or drug dependence or abuse. If the subject has a recent history of substance abuse, there will be a two-week washout period before initiating the trial as an added precaution. There are no known safety issues relating to memantine and recent history of substance abuse.
* Serious, stable or unstable systemic illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
* Subjects with severe hepatic impairment (LFTs > 3 times ULN).
* Subjects with genitourinary conditions that raise urine pH (e.g., renal tubular acidosis, severe infection of the urinary tract).
* Known hypersensitivity to memantine.
* Severe allergies or multiple adverse drug reactions.
* A history of intolerance or adequate exposure to memantine, as determined by the clinician.
* Investigator and his/her immediate family defined as the investigator's spouse, parent, child, grandparent, or grandchild.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression-Improvement Scale (CGI-I) | Baseline to 12 weeks
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale (1 to 7-- with higher numbers indicating more severely affected) that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Brignell A, Marraffa C, Williams K, May T. Memantine for autism spectrum disorder. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013845. doi: 10.1002/14651858.CD013845.pub2. PMID 36006807